CLINICAL TRIAL: NCT07106606
Title: The Effect of the Mandala Method in Reduction of Psychological Distress During Anogenital Examination of Sexually Abused Children Aged 9-12
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Nurgül Bozkurt, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022/107
Record Dates: First submitted 2025-07-22; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Anxiety; Sexual Abuse of Child (If Focus of Attention is on Victim); Fear and Anxiety
Keywords: anogenital examination; Sexual abuse of child; Child Monitoring Center; Mandala; anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Comparator (Active Comparator): The group completed a structured mandala-coloring activity prior to the examination.
  Interventions: Behavioral: Mandala coloring activity
- Control group (No Intervention): The group only received routine information before the examination.

INTERVENTIONS:
Behavioral: Mandala coloring activity — This technique is a creative art-based relaxation method that aims to reduce children's anxiety and fear levels. The application was carried out to make children feel psychologically safer and calmer before the examination. The selected mandala forms were created in accordance with the attention span, motor skill capacity and visual perception development of children between the ages of 9 and 12 by choosing simple but symbolic structures with moderate level of detail.
  Arms: Active Comparator

SUMMARY:
The goal of this study is evaluating the effectiveness of a mandala-coloring intervention in reducing psychological distress (fear, state anxiety, and related physiological indicators) during anogenital examinations among sexually abused children aged 9-12.

ELIGIBILITY:
Inclusion Criteria:

* Coming to anogenital examination for the first time,
* The child and parents have native Turkish language skills and the ability to read and write.

Exclusion Criteria:

* Sensory loss at a level that prevents communication with the child,
* Intelligence quotient (IQ) of 55 and below in the records,
* Has a mental or neurological disability that prevents communication.

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 68 (Actual)
Dates: Start 2024-05-10 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-06-03 (Actual)

PRIMARY OUTCOMES:
Findings on Anxiety Level | Baseline, half an hour before the anogenital examination and immediately after anogenital examination
  State Anxiety Inventory for Children used in this study. It was developed by Spielberger to measure state and trait anxiety levels of children aged 9-12 years. Its adaptation into Turkish, validity and reliability study was conducted by Özusta (1993). It consists of two subscales, "state anxiety" and "trait anxiety", each consisting of 20 items.
  State anxiety subscale: Measures how the child feels "at that moment". Trait anxiety subscale: Measures how the child feels "in general". Both subscales give scores ranging from 20 to 60. In this study, since the change in state anxiety level before and after the anogenital examination will be evaluated, the "state anxiety" subscale was predominantly reflected in the findings. However, although trait anxiety was not examined in pre- and post-examination comparison, this subscale was also examined in the pre-test and post-test measurements. The Cronbach's alpha coefficient of state anxiety subscale was 0.82 and trait anxiety subscale was 0.81
Findings on Fear Level | Baseline, half an hour before the anogenital examination and immediately after anogenital examination
  Children's Fear Scale: It is a single-item scale consisting of 5 facial expressions. The first facial expression is scored as neutral (0) and the last facial expression as the highest fear (4). It is used to measure the fear level of children before and after the procedure (blood sampling, examination, etc.) (McMurtry et al., 2011). In this study, it was used to determine the change in fear level before and after anogenital examination. Since it includes a single scoring, the reliability coefficient was not calculated.

SECONDARY OUTCOMES:
Cardiac Pulse Finding | Baseline, half an hour before the anogenital examination and immediately after anogenital examination
  It is a form in which the pulse (beats/min) counts and the scores obtained from the scales are recorded before and after the examination.
Respiratory Rate Finding | Baseline, half an hour before the anogenital examination and immediately after anogenital examination
  It is a form in which the respiration (breaths/min) counts and the scores obtained from the scales are recorded before and after the examination.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Basaksehir Cam and Sakura City Hospital Child Advocacy Center, Istanbul, Basaksehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available on request
Supporting Information: Study Protocol, SAP, ICF